CLINICAL TRIAL: NCT01158833
Title: Validity of the Kinematic Classification of Gait in Diplegic Children With Cerebral Palsy
Brief Title: Validity of the Kinematic Classification of Gait in Diplegic Children With Cerebral Palsy (CP)
Status: Completed | Type: Observational
Sponsor: University of Modena and Reggio Emilia (Other)
Collaborators: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Principal Investigator, Stefania Costi, Physical Therapist, University of Modena and Reggio Emilia
Other Study IDs: UDGEE_2010_classdipl
Record Dates: First submitted 2010-07-06; First posted 2010-07-08 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Cerebral Palsy; Diplegia, Spastic
Keywords: Cerebral palsy; diplegia; gait; classification
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- spastic diplegia due to Cerebral Palsy
  Interventions: Other: classification of gait in diplegic children with CP

INTERVENTIONS:
Other: classification of gait in diplegic children with CP — To determine the criterion validity of the classification of the pattern of diplegic gait proposed by Ferrari et al. we correlated gait patterns with the score of the FMS.

SUMMARY:
In recent years Ferrari et al. proposed a new classification of gait in diplegic children with spastic diplegia that describes four different patterns of gait by analyzing the strategies that each children adopts to need his/her needs to walk. The investigators believe that this classification provides the clinician with clinically meaningful information in terms of coping strategies adopted to maximize the ability to walk.

The aim of this study is to determine the criterion validity of the new classification of the pattern of gait in children with spastic diplegia by correlating pattern of diplegic gait with the score of the Functional performance measure.

ELIGIBILITY:
Inclusion Criteria:

* diplegia and CP;

Exclusion Criteria:

* severe mental retardation attested by the Diagnostic and Statistical Manual of mental disorders IV
* pharmaco-resistant epilepsy
* behavioural disorders

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We retrospectively studied children with diplegia and CP who are followed by the Unit for Severe Disability in the Developmental Age at the Hospital of Reggio Emilia (Italy);
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Functional Mobility Scale (FMS) | at the age of 12 to 17 years
  correlation between the new classification of diplegic gait and the FMS which classifies the functional mobility in children

CONTACTS AND LOCATIONS:
Overall Officials: Adriano Ferrari, MD, Study Chair — University of Modena and Reggio Emilia and Hospital Santa Maria Nuova; Stefania Costi, PT, Study Director — University of Modena and Reggio Emilia; Rita Neviani, PT, Principal Investigator — Azienda USL Reggio Emilia - IRCCS
Locations (1):
- Arcispedale Santa Maria Nuova, Reggio Emilia, RE, Italy

REFERENCES:
- [Background] Pascale R, Perazza S, Borelli G, Bianchini E, Alboresi S, Paolicelli PB, Ferrari A, Cioni G. The term diplegia should be enhanced. Part III: inter-observer reliability of the new rehabilitation oriented classification. Eur J Phys Rehabil Med. 2008 Jun;44(2):213-20. PMID 18418341
- [Background] Cioni G, Lodesani M, Pascale R, Coluccini M, Sassi S, Paolicelli PB, Perazza S, Ferrari A. The term diplegia should be enhanced. Part II: contribution to validation of the new rehabilitation oriented classification. Eur J Phys Rehabil Med. 2008 Jun;44(2):203-11. PMID 18418340
- [Background] Ferrari A, Alboresi S, Muzzini S, Pascale R, Perazza S, Cioni G. The term diplegia should be enhanced. Part I: a new rehabilitation oriented classification of cerebral palsy. Eur J Phys Rehabil Med. 2008 Jun;44(2):195-201. PMID 18418339